CLINICAL TRIAL: NCT05958134
Title: Brazilian Reality in the Diagnosis and Treatment of Diffuse Large B Cell Lymphoma - BRA-DLBCL: Multicenter Retrospective Study (Real World Evidence - RWE)
Brief Title: Brazilian Reality in the Diagnosis and Treatment of Diffuse Large B Cell Lymphoma - BRA-DLBCL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: D133HR00022; BRA-DLBCL (Other: Hospital Israelita Albert Einstein)
Record Dates: First submitted 2023-07-04; First posted 2023-07-24 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Lymphoma; RWE; Diffuse Large B Cell
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnosed with diffuse large B-cell lymphoma, and classified regarding the cell of origin: Retrospective data collection will be carried out from the medical records of the participants included in the study. Will be held description of the epidemiological profile and pathological staging of diffuse large B-cell lymphoma conditions (DLBCL/LDGCB), imaging profiling, together with first-line treatment used in subgroups of germinal center or activated B-cell, in patients followed in Brazilian reference cancer treatment centers, within the last 6 years (between 2017 and 2022).

SUMMARY:
National, multicenter, non-randomized, retrospective observational study (Real World Evidence-RWE) to analyze the epidemiological profile of diffuse large B cell lymphoma, clinical management, treatment in molecular subgroups, progression profile and patient survival outcomes enrolled and treated within the last 6 years (2017 to 2022), in national cancer reference centers.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma management is a challenge in clinical setting, as the heterogeneity of conditions due to the molecular complexity of DLBCL may limit treatment response. Other major factor is that in Brazil we lack evidence of treatment response profiling regarding this molecular complexity. To know the epidemiological profile of DLBCL, together with the first-line treatment profile that has been adopted in reference centers, as well as the management of relapsing, is essentially important in generating evidence that add up to actions targeting the improvement of patient care, providing them with better treatments. The Brazilian reality of clinical presentation, management profile, employed treatments and response rate is little known. Considering the Brazilian reality of a continental country, where healthcare services in reference centers present heterogeneous realities, analyzing clinical routine data may generate important evidence (RWE) to comprise the understanding on treatments effectiveness. Generated evidence has the potential to help understanding the reality of Brazilian patients, as well as supporting new regional researches.

ELIGIBILITY:
Inclusion Criteria:

* Male and female;
* Age above 18 years old;
* Diagnosis of diffuse large B-cell lymphoma (DLBCL) and high-grade non-Hodgkin B-cell lymphoma at all stagings;
* Lymphoma classified for the cell of origin (GCB - Germinal Center B-Cell lymphoma, and non-germinal center);
* Having first life of treatment information available in institutional medical record;
* Having survival data available in institutional medical record.

Exclusion Criteria:

* No medical record of the molecular subgroup classification;
* Diagnosis of diffuse large B-cell lymphoma, confirmed in the year 2016;
* Patients diagnosed with Transformed Lymphomas.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with diffuse large B-cell lymphoma, who meet the eligibility criteria and have been treated and followed in the study participating sites within the last 6 years (from 2017 to 2022) will be included in the study.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Disease staging | Time Frame: 6 years (Time of retrospective observational analysis of the study)
  Description of the staging of diffuse large B-cell lymphoma conditions in patients followed in Brazilian reference cancer treatment centers
Time between diagnosis and start of treatment | Time Frame: 6 years (Time of retrospective observational analysis of the study)
  Description of the time between diagnosis and start of treatment
Progression-free Survival | Time Frame: 6 years (Time of retrospective observational analysis of the study)
  Progression-free Survival will be evaluated as the time from the beginning of treatment, considering each line of treatment, to the objective progression of tumor or death
Overall Survival | Time Frame: 6 years (Time of retrospective observational analysis of the study)
  Overall Survival will be evaluated as the time from the diagnosis of the hematological disease at any staging until all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Fleury Perini, Principal Investigator — Hospital Israelita Albert Einstein
Locations (4):
- Brazil (4):
  - Research Site, Belo Horizonte
  - Research Site, Recife
  - Research Site, Salvador
  - Research Site, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133HR00022&attachmentIdentifier=d59beb8c-91f2-4987-b727-9e0f737a01d3&fileName=D133HR00022_Clinical_Study_Report_Synopsis.pdf&versionIdentifier=